CLINICAL TRIAL: NCT00001000
Title: Immunologic Effect After Single Dose Atvogen in Healthy Volunteers and Asymptomatic HIV-Infected Patients
Brief Title: A Study of Atvogen in Healthy Volunteers and HIV-Infected Patients Who Have No Symptoms of Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Masking: Double | Purpose: Treatment
Other Study IDs: ACTG 056; 11030 (Registry Identifier: DAIDS-ES)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2012-10-19 (Estimated); Status verified 2012-10

CONDITIONS: HIV Infections
Keywords: Macrophage Activation; Lymphocyte Transformation; Immunologic Surveillance; ampligen; Antiviral Agents
MeSH Terms: conditions — HIV Infections | interventions — poly(I).poly(c12,U)

INTERVENTIONS:
Drug: Ampligen

SUMMARY:
To evaluate the degree and sequence of immunologic enhancement and the cellular resistance to certain infections after a single dose of atvogen (ampligen). In addition, the relationship between activation of immune cells and biochemical markers of that activation will be studied.

Treatment of patients with HIV infection must address both the primary viral infection and the subsequent immune deficiency, which is the primary cause of mortality in AIDS. In vitro studies of ampligen have shown it will inhibit HIV infection. Ampligen may also minimize the toxicity of many drugs used in the treatment of AIDS and induce an antiviral state in the brain that may be useful in treating neurologic symptoms of HIV infection. The time course and degree of immunologic response to ampligen remain unknown although they are essential for proper use of the drug in the treatment of HIV infection and perhaps other clinical problems.

DETAILED DESCRIPTION:
Treatment of patients with HIV infection must address both the primary viral infection and the subsequent immune deficiency, which is the primary cause of mortality in AIDS. In vitro studies of ampligen have shown it will inhibit HIV infection. Ampligen may also minimize the toxicity of many drugs used in the treatment of AIDS and induce an antiviral state in the brain that may be useful in treating neurologic symptoms of HIV infection. The time course and degree of immunologic response to ampligen remain unknown although they are essential for proper use of the drug in the treatment of HIV infection and perhaps other clinical problems.

Ten healthy volunteers and 10 HIV-infected patients are randomized between ampligen or placebo group. Five volunteers in each group receive a single dose of ampligen on day 1 and a single dose of placebo on day 8. The other 5 volunteers receive the drug and placebo on day 8 and 1, respectively. Seven days of observation and testing follow each administration of drug or placebo and also allow the body to eliminate the drug.

ELIGIBILITY:
Inclusion Criteria

Patients' general good health should be determined by screening history, physical examination, and laboratory tests including CBC with differential, erythrocyte sedimentation rate, urinalysis, SMA-24, and drug screen within the established limits of normal for the hospital laboratory.

Exclusion Criteria

Co-existing Condition:

The following subjects will be excluded from the study:

* Smokers.
* Volunteers who have ingested alcohol 48 hours prior to the study.
* Volunteers with clinically apparent viral disease or other illnesses, including allergies, within 2 weeks prior to the study or conditions which predispose them to chronic immune stimulation.

Concurrent Medication:

Excluded:

* All medications.

The following subjects will be excluded from the study:

* Smokers.
* Volunteers who have ingested alcohol 48 hours prior to the study.
* Volunteers with clinically apparent viral disease or other illnesses, including allergies, within 2 weeks prior to the study or conditions which predispose them to chronic immune stimulation.

Prior Medication:

Excluded within 2 weeks of study entry:

* All medications.

Recent history of drug or alcohol abuse.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20
Dates: Study Completion 1990-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: PS Lietman, Study Chair
Locations (1):
- Johns Hopkins Hosp, Baltimore, Maryland, United States

REFERENCES:
- [Background] Hendrix CW, Margolick JB, Petty BG, Markham RB, Nerhood L, Farzadegan H, Ts'o PO, Lietman PS. Biologic effects after a single dose of poly(I):poly(C12U) in healthy volunteers. Antimicrob Agents Chemother. 1993 Mar;37(3):429-35. doi: 10.1128/AAC.37.3.429. PMID 7681656